CLINICAL TRIAL: NCT00004838
Title: Randomized Study of Succimer (Dimercaptosuccinic Acid) on Growth of Lead-Poisoned Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Nationwide Children's Hospital (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13576; CHRF-96-HS-066; CH-OHIO-5F32ES05651
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-09

CONDITIONS: Lead Poisoning
Keywords: environmental/toxic disorders; lead poisoning; rare disease
MeSH Terms: conditions — Lead Poisoning; Rare Diseases | interventions — Succimer

INTERVENTIONS:
Drug: succimer

SUMMARY:
OBJECTIVES:

Compare growth of lead-poisoned children receiving succimer (dimercaptosuccinic acid; DMSA) plus standard treatment to those receiving standard treatment only.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is randomized study. Patients are randomized to receive succimer in addition to standard treatment (arm I) or standard treatment only (arm II).

Succimer is administered orally 3 times a day for 7 days, then twice daily for 19 days. Patients may receive up to 3 courses.

Standard treatment consists of a medical history and physical examination, environmental assessment with modification to reduce lead exposure, dietary modifications to decrease lead absorption, the use of a daily multivitamin and mineral supplement with iron, developmental screening and intervention, and frequent follow up of lead levels.

If blood lead level rises above 45 mcg/dL, patient receives succimer regardless of treatment arm originally assigned.

Patients are followed every 3-4 weeks for 2 months, then every 3 months for 6 months, and then every 6 months thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Asymptomatic children with confirmed venous blood lead of at least 20 mcg/dL and less than 45 mcg/dL Children with blood lead of 45 mcg/dL or greater are not randomized in this study since they probably will receive succimer regardless of being enrolled in this study --Patient Characteristics-- Other: No contraindications to the use of succimer (i.e., allergy or a lack of lead safe environment in which to live during chelation)

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175
Dates: Start 1997-09; Study Completion 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Marcel J. Casavant, Study Chair — Nationwide Children's Hospital

REFERENCES:
- [Background] The Treatment of Lead-exposed Children (TLC) trial: design and recruitment for a study of the effect of oral chelation on growth and development in toddlers. Paediatr Perinat Epidemiol. 1998 Jul;12(3):313-33. doi: 10.1046/j.1365-3016.1998.00122.x. PMID 9690266